CLINICAL TRIAL: NCT03499899
Title: A Phase II Open-label, Randomized, Three-arm, Multicenter Study of LAG525 Given in Combination With Spartalizumab (PDR001), or With Spartalizumab and Carboplatin, or With Carboplatin, as First or Second Line Therapy in Patients With Advanced Triple-negative Breast Cancer
Brief Title: A Study of Efficacy and Safety of LAG525 in Combination With Spartalizumab, or With Spartalizumab and Carboplatin, or With Carboplatin, in Patients With Advanced Triple-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAG525B2101; 2017-004865-28 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-17 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Triple-negative Breast Cancer
Keywords: advanced triple-negative breast cancer; triple-negative breast cancer; checkpoint inhibition; LAG525; spartalizumab; PDR001; carboplatin
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — spartalizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LAG525 + PDR001 (Experimental): Participants received LAG525 and PDR001 administered as infusion once every 3 weeks
  Interventions: Drug: LAG525; Drug: PDR001
- LAG525 + PDR001 + carboplatin (Experimental): Participants received LAG525, PDR001 and carboplatin administered as infusion once every 3 weeks.
  Interventions: Drug: LAG525; Drug: PDR001; Drug: Carboplatin
- LAG525 + carboplatin (Experimental): Participants received LAG525 and carboplatin administered as infusion once every 3 weeks
  Interventions: Drug: LAG525; Drug: Carboplatin

INTERVENTIONS:
Drug: LAG525 — LAG525 was a concentrate for solution for intravenous infusion, came in 100mg vials as a liquid formulation for infusion and was dosed at 400mg every 21 days. For all arms, LAG525 was infused first
Drug: PDR001 — Spartalizumab was a concentrate for solution for intravenous infusion, came in 100mg vials as a liquid formulation for infusion and was dosed at 300mg every 21 days. Spartalizumab was infused after LAG525
  Other Names: Spartalizumab
  Arms: LAG525 + PDR001; LAG525 + PDR001 + carboplatin
Drug: Carboplatin — Carboplatin was a concentrate for solution for intravenous infusion, came in 100mg/mL and was dosed per area under the curve (AUC) 6 every 21 days. Carboplatin was infused once LAG525 and spartalizumab infusions were completed
  Arms: LAG525 + PDR001 + carboplatin; LAG525 + carboplatin

SUMMARY:
The main purpose of this study was to assess the antitumor activity of three combinations: i) LAG525 + spartalizumab; ii) LAG525 + spartalizumab + carboplatin, and iii) LAG525 + carboplatin in participants with advanced triple-negative breast cancer (TNBC) in first or second line therapy.

DETAILED DESCRIPTION:
This was an open-label, Phase II, randomized, multicenter study to assess the efficacy, safety, and pharmacokinetic characteristics of the following three combinations: LAG525 + spartalizumab (PDR001) (Arm 1), LAG525 + spartalizumab (PDR001) + carboplatin (Arm 2), and LAG525 + carboplatin (Arm 3) in participants with advanced triple-negative breast cancer (TNBC) which progressed after adjuvant or one prior line of systemic therapy for metastatic disease.

Participants were assigned to one of the three treatment arms in a ratio of 1:1:1. In protocol amendment 3 (released on 28-Mar-2019), enrollment to treatment Arm 1 (LAG525 + spartalizumab) was prematurely closed due to a higher discontinuation rate due to progressive disease and all subsequent enrolled patients were randomized to Arms 2 and 3 only, in a ratio of 1:1.

Study treatment continued until disease progression, unacceptable toxicity, pregnancy, investigator/participant decision, start of a new anti-neoplastic therapy, withdrawal of consent, lost to follow-up, death, or study was terminated by the sponsor. The investigator might decide to stop carboplatin after 6 cycles, even if the above criteria were not met. Participants who continued to derive clinical benefit from the treatment based on the investigator's evaluation following their completion of this trial might receive post-trial access (PTA) i.e. rollover protocol or a post-study drug supply (PSDS).

The end of study was defined as the earliest occurrence of one of the following: (1) all participants had died or (2) discontinued from the study, or (3) another clinical study became available that could continue to provide study treatment in this participant population and all ongoing participants were eligible to be transferred to that clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Had advanced (loco-regionally recurrent not amenable to curative therapy or metastatic) breast cancer
* Had adequate bone marrow and organ function.
* Had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Had measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria (Tumor lesions previously irradiated or subjected to other loco-regional therapy was to be considered measurable if disease progression at the treated site after completion of therapy is clearly documented)
* Progressed after adjuvant or 1 prior systemic treatment in the metastatic setting. Patients with de novo metastatic disease were eligible if they received 1 prior line of therapy
* Had received prior systemic treatment that included taxane-based chemotherapy for adjuvant or metastatic disease
* Had a site of disease amenable to biopsy, and was willing to undergo a new tumor biopsy at screening and during therapy on this study, the latter if medically feasible. Patients with an available archival tumor tissue did not need to perform a tumor biopsy at screening if patient had not received anti-cancer therapy since the biopsy was taken.
* Had histologically and/or cytologically confirmed diagnosis of advanced TNBC (based on most recently analyzed biopsy from locally recurrent or metastatic site, local lab) meeting the following criteria: HER2 negative in situ hybridization test or an IHC status of 0 or 1+, and ER and PR expression was <1 percent as determined by immunohistochemistry (IHC)

Exclusion Criteria:

* Had received prior immune checkpoint inhibitors as anticancer treatment such as anti-LAG-3, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody (any line of therapy)
* Received prior neoadjuvant or adjuvant therapy with a platinum agent or mitomycin and experienced recurrence within 12 months after the end of the platinum-based or mitomycin containing therapy or received Platinum or mitomycin for metastatic disease
* Had major surgery within 14 days prior to starting study treatment or had not recovered to grade 1 or less from major side effects
* Presence of CTCAE grade 2 toxicity or higher due to prior cancer therapy. Exception to this criterion; patients with any grade of alopecia were allowed to enter the study.
* Had received radiotherapy ≤ 4 weeks prior to randomization (≤ 2 weeks for limited field radiation for palliation), and had not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia)
* Had a known hypersensitivity to other monoclonal antibodies, platinum-containing compounds, or to any of the excipients of LAG525, spartalizumab, or carboplatin
* Had symptomatic central nervous system (CNS) metastases or CNS metastases that required local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within the 2 weeks prior to first dose of study treatment. Patients with treated brain metastases would be neurologically stable and without CNS progression for at least 12 weeks prior to randomization and had discontinued corticosteroid treatment (with the exception of < 10 mg/day of prednisone or equivalent for an indication other than CNS metastases) for at least 4 weeks before first dose of any study treatment
* Had clinically significant cardiac disease or impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (2):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Australia (3):
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Novartis Investigative Site, Liège, Belgium
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec
- Novartis Investigative Site, Paris, France
- Germany (3):
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Tübingen
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Napoli, Italy
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Minato Ku, Tokyo
- Lebanon (3):
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, El Metn
  - Novartis Investigative Site, Saida
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 33 centers in 17 countries.
Pre-assignment Details: A total of 132 participants were screened of which 88 participants were enrolled in the study and 87 participants received at least one dose of study treatment (1 participant was not treated due to physician decision)
Groups:
- LAG525+ PDR001+ Carboplatin: Participants received LAG525, PDR001 and carboplatin administered as infusion once every 3 weeks.
Period: Overall Study
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Started | 20 | 34 | 34
Treated | 19 | 34 | 34
Completed | 0 | 0 | 0
Not Completed | 20 | 34 | 34
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 3 | 6 | 6
Not completed — Progressive disease | 15 | 23 | 23
Not completed — Patient decision | 0 | 1 | 1
Not completed — Terminated by sponsor (end of study definition was met) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin | Total
Number analyzed (Participants) | 20 | 34 | 34 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (10.22) | 50.9 (10.88) | 53.3 (10.78) | 52.5 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 34 | 34 | 88
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 8 | 7 | 23
  Black or African American | 0 | 0 | 1 | 1
  Missing | 0 | 3 | 1 | 4
  White | 12 | 23 | 25 | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Investigator's Assessment According to RECIST v1.1
Description: Overall response rate (ORR) is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 based on investigator's assessment. The 95% CIs were computed using two-sided exact binomial method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 14 months
Population: Full Analysis Set (FAS): All participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 20 | 34 | 34
Percentage of participants | 5.0 [0.1 to 24.9] | 32.4 [17.4 to 50.5] | 17.6 [6.8 to 34.5]

2. Secondary Outcome: Clinical Benefit Rate (CBR) Per Investigator's Assessment According to RECIST v1.1
Description: CBR is defined as the percentage of participants with a best overall response (BOR) of confirmed CR or PR, or stable disease (SD) lasting 24 weeks or longer, according to RECIST 1.1 criteria. The 95% CI were computed using two-sided exact binomial method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 14 months
Population: FAS: All participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 20 | 34 | 34
Percentage of Participants | 5.0 [0.1 to 24.9] | 35.3 [19.7 to 53.5] | 20.6 [8.7 to 37.9]

3. Secondary Outcome: Duration of Response (DOR) Per Investigator's Assessment According to RECIST v1.1
Description: DOR is the time between the first documented response (CR or PR) and the first documented progression or death due to underlying cancer based on RECIST1.1 and as per investigator's assessment. The DOR distribution was estimated using the Kaplan-Meier method and the 95% confidence intervals using the method of Brookmeyer and Crowley. If progression or death did not occur, the participant was censored at the date of last adequate tumor assessment.
  CR: Disappearance of all non-nodal target lesions and any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  Progression: at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first documented response up to disease progression or death due to underlying cancer, whichever occurs first, up to approximately 14 months
Population: Participants with a confirmed CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 1 | 11 | 6
Months | 4.9 [NA to NA] — NA: Confidence Interval was not estimable due to the low number of events | 13.6 [2.8 to NA] — NA: Upper limit of the confidence Intervals was not estimable due to the low number of events | 12.6 [2.4 to NA] — NA: Upper limit of the confidence Intervals was not estimable due to the low number of events

4. Secondary Outcome: Time to Response (TTR) Per Investigator's Assessment According to RECIST v1.1
Description: TTR is the time from date of randomization to first documented response of CR or PR based on investigators' assessment and according to RECIST 1.1. Median TTR was summarized using descriptive statistics.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of randomization to first documented response (CR or PR), up to approximately 14 months
Population: Participants with a confirmed CR or PR
Measure: Median (Full Range); unit: Months
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 1 | 11 | 6
Months | 1.5 [1.5 to 1.5] | 1.7 [1.2 to 4.1] | 1.4 [1.2 to 2.8]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time from date of randomization to the date of first documented progression or death due to any cause. PFS was assessed via investigator's assessment according to RECIST 1.1. PFS was censored at the date of the last adequate tumor assessment if no PFS event was observed prior to the analysis cut-off date or before the start of the new anticancer therapy date, whichever is earlier. The PFS distribution was estimated using the Kaplan-Meier method. The 95% confidence intervals were calculated using the method of Brookmeyer and Crowley.
Time Frame: From date of randomization to disease progression or death due to any cause, whichever occurs first, up to approximately 14 months
Population: FAS: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 20 | 34 | 34
Months | 1.4 [1.2 to 1.5] | 4.3 [2.8 to 5.6] | 3.0 [2.2 to 5.5]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death due to any cause. If a participant was not known to have died, then OS was censored at the latest date the participant was known to be alive (on or before the cut-off date). The OS distribution was estimated using the Kaplan-Meier method. The 95% confidence intervals were calculated using the method of Brookmeyer and Crowley
Time Frame: From date of randomization to date of death due to any cause, up to 18 months
Population: FAS: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 20 | 34 | 34
Months | 6.1 [4.6 to NA] — NA: Upper limit of the confidence interval was not estimable due to the low number of events | 11.6 [7.5 to NA] — NA: Upper limit of the confidence interval was not estimable due to the low number of events | 8.0 [6.2 to 9.3]

7. Secondary Outcome: Pharmacokinetics (PK) Parameter, Area Under the Plasma Concentration Versus Time Curve From Time 0 to 504 Hours (AUC0-504h) of LAG525
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUC0-504h was defined as the area under the plasma concentration-time curve from time zero to 504h.
Time Frame: Cycle 1 at pre-infusion, 1 hour (hr) post end of infusion, 168 hr, 336 hr and 504 hr post-infusion on Day 1 of Cycle 1. Cycle 3 at pre-infusion, 1 hr post end of infusion, 168 hr, 336 hr and 504 hr post-infusion on Day 1 of Cycle 3. Each cycle is 21 days
Population: LAG525 pharmacokinetic analysis set (PAS-LAG525) including all participants who provided at least one evaluable LAG525 PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram/miliLiter (day*ug/mL)
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 11 | 24 | 33
day*microgram/miliLiter (day*ug/mL)
  Cycle 1: number analyzed (Participants) | 11 | 19 | 22
  Cycle 1 | 1270 (25.8) | 1350 (22.4) | 1180 (23.4)
  Cycle 3: number analyzed (Participants) | 3 | 14 | 11
  Cycle 3 | 2060 (60.1) | 2200 (34.4) | 1990 (31.3)

8. Secondary Outcome: PK Parameter, Cmax of LAG525
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Cmax is the maximum observed plasma LAG525 concentration
Time Frame: as for outcome 7
Population: PAS-LAG525 including all participants who provided at least one evaluable LAG525 PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 16 | 34 | 30
ug/mL
  Cycle 1: number analyzed (Participants) | 16 | 31 | 28
  Cycle 1 | 127 (26.5) | 136 (21.1) | 128 (17.9)
  Cycle 3: number analyzed (Participants) | 6 | 23 | 24
  Cycle 3 | 144 (48.9) | 181 (29.5) | 168 (26.6)

9. Secondary Outcome: PK Parameter, AUClast of LAG525
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast) of LAG525
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 16 | 34 | 29
day*ug/mL
  Cycle 1: number analyzed (Participants) | 16 | 31 | 28
  Cycle 1 | 1170 (32.0) | 1310 (41.1) | 1010 (151.2)
  Cycle 3: number analyzed (Participants) | 6 | 23 | 24
  Cycle 3 | 240 (9775.4) | 2040 (49.8) | 1490 (196.4)

10. Secondary Outcome: PK Parameter, Tmax of LAG525
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Tmax is the time to reach maximum LAG525 serum concentration. Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 16 | 34 | 30
hr
  Cycle 1: number analyzed (Participants) | 16 | 31 | 28
  Cycle 1 | 1.51 (40.7) | 1.76 (35.5) | 1.58 (23.1)
  Cycle 3: number analyzed (Participants) | 6 | 23 | 24
  Cycle 3 | 1.64 (13.4) | 1.58 (15.0) | 1.77 (37.4)

11. Secondary Outcome: PK Parameter, AUC0-504h of PDR001
Description: as for outcome 7
Time Frame: as for outcome 7
Population: PDR001 pharmacokinetic analysis set (PAS-PDR001) including all participants who provided at least one evaluable PDR001 PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 11 | 24
day*ug/mL
  Cycle 1: number analyzed (Participants) | 11 | 18
  Cycle 1 | 819 (23.6) | 907 (29.1)
  Cycle 3: number analyzed (Participants) | 3 | 15
  Cycle 3 | 1490 (41.0) | 1710 (29.5)

12. Secondary Outcome: PK Parameter, Cmax of PDR001
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Cmax is the maximum observed PDR001 serum concentration
Time Frame: as for outcome 7
Population: PAS-PDR001 including all participants who provided at least one evaluable PDR001 PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 16 | 33
ug/mL
  Cycle 1: number analyzed (Participants) | 16 | 28
  Cycle 1 | 78.0 (18.9) | 82.4 (25.1)
  Cycle 3: number analyzed (Participants) | 6 | 21
  Cycle 3 | 95.1 (41.4) | 117 (26.8)

13. Secondary Outcome: PK Parameter, AUClast of PDR001
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast) of PDR001
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 16 | 33
day*ug/mL
  Cycle 1: number analyzed (Participants) | 16 | 28
  Cycle 1 | 780 (24.4) | 890 (44.6)
  Cycle 3: number analyzed (Participants) | 5 | 21
  Cycle 3 | 374 (2703.2) | 1500 (55.7)

14. Secondary Outcome: PK Parameter, Tmax of PDR001
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Tmax is the time to reach maximum PDR001 serum concentration. Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 16 | 33
hr
  Cycle 1: number analyzed (Participants) | 16 | 28
  Cycle 1 | 1.43 (34.7) | 1.71 (29.7)
  Cycle 3: number analyzed (Participants) | 6 | 21
  Cycle 3 | 1.67 (13.6) | 1.61 (13.9)

15. Secondary Outcome: PK Parameter, AUC0-4h of Carboplatin (Total Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUC0-4h was defined as the area under the plasma concentration-time curve from time zero to 4h (determined as total platinum).
Time Frame: Cycle 1 at pre-infusion, end of infusion, 1 hour, 2 hours and 3 hours post end of infusion. Cycle 3 at pre-infusion, end of infusion, 1 hour, 2 hours and 3 hours post end of infusion. Each cycle is 21 days
Population: Carboplatin (plasma) PAS including all participants who provided at least one evaluable carboplatin PK plasma concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/miliLiter (hr*ng/mL)
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 24 | 20
hour*nanogram/miliLiter (hr*ng/mL)
  Cycle 1: number analyzed (Participants) | 20 | 16
  Cycle 1 | 45000 (23.0) | 45200 (16.1)
  Cycle 3: number analyzed (Participants) | 14 | 14
  Cycle 3 | 42700 (27.6) | 43500 (29.2)

16. Secondary Outcome: PK Parameter, Cmax of Carboplatin (Total Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Cmax is the maximum observed carboplatin plasma concentration (determined as total platinum)
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 33 | 31
ng/mL
  Cycle 1: number analyzed (Participants) | 30 | 27
  Cycle 1 | 22300 (32.0) | 21400 (32.2)
  Cycle 3: number analyzed (Participants) | 23 | 23
  Cycle 3 | 20900 (33.4) | 20000 (199.2)

17. Secondary Outcome: PK Parameter, AUClast of Carboplatin (Total Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast) of carboplatin (determined as total platinum)
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 33 | 29
ng/mL
  Cycle 1: number analyzed (Participants) | 28 | 25
  Cycle 1 | 42000 (30.8) | 38900 (56.3)
  Cycle 3: number analyzed (Participants) | 23 | 22
  Cycle 3 | 40800 (38.1) | 42600 (43.3)

18. Secondary Outcome: PK Parameter, Tmax of Carboplatin (Total Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Tmax is the time to reach maximum carboplatin plasma concentration (determined as total platinum). Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 15
Population: Carboplatin (plasma) PAS including all participants who provided at least one evaluable carboplatin PK plasma concentration.Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 33 | 31
hr
  Cycle 1: number analyzed (Participants) | 30 | 27
  Cycle 1 | 0.857 (35.5) | 0.720 (31.9)
  Cycle 3: number analyzed (Participants) | 23 | 23
  Cycle 3 | 0.789 (33.0) | 0.720 (34.8)

19. Secondary Outcome: PK Parameter, AUC0-4h of Carboplatin (Ultrafilterable Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUC0-4h was defined as the area under the plasma concentration-time curve from time zero to 4h (determined as ultrafilterable platinum).
Time Frame: as for outcome 15
Population: Carboplatin (plasma ultrafiltrate) PAS including all participants who provided at least one evaluable carboplatin PK plasma ultrafiltrate concentration. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/miliLiter (hr*ng/mL)
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 12 | 7
hour*nanogram/miliLiter (hr*ng/mL)
  Cycle 1: number analyzed (Participants) | 8 | 5
  Cycle 1 | 43600 (13.1) | 44700 (23.4)
  Cycle 3: number analyzed (Participants) | 9 | 5
  Cycle 3 | 41100 (30.5) | 41000 (12.8)

20. Secondary Outcome: PK Parameter, Cmax of Carboplatin (Ultrafilterable Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Cmax is the maximum observed carboplatin plasma concentration (determined as ultrafilterable platinum)
Time Frame: as for outcome 15
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 15 | 19
ng/mL
  Cycle 1: number analyzed (Participants) | 12 | 13
  Cycle 1 | 23200 (19.8) | 25700 (24.2)
  Cycle 3: number analyzed (Participants) | 12 | 12
  Cycle 3 | 22300 (40.1) | 14700 (4159.6)

21. Secondary Outcome: PK Parameter, AUClast of Carboplatin (Ultrafilterable Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. AUClast is the area under the curve (AUC) from time zero to the last measurable concentration sampling time (tlast) of carboplatin (determined as ultrafilterable platinum)
Time Frame: as for outcome 15
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 15 | 17
ng/mL
  Cycle 1: number analyzed (Participants) | 10 | 11
  Cycle 1 | 41400 (13.0) | 35600 (65.2)
  Cycle 3: number analyzed (Participants) | 12 | 11
  Cycle 3 | 37400 (30.1) | 36300 (68.2)

22. Secondary Outcome: PK Parameter, Tmax of Carboplatin (Ultrafilterable Platinum)
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Tmax is the time to reach maximum carboplatin plasma concentration (determined as ultrafilterable platinum). Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 15
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 15 | 19
hr
  Cycle 1: number analyzed (Participants) | 12 | 13
  Cycle 1 | 0.802 (42.5) | 0.660 (34.4)
  Cycle 3: number analyzed (Participants) | 12 | 12
  Cycle 3 | 0.828 (39.7) | 0.686 (34.6)

23. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) at Baseline for LAG525
Description: Number of participants who had an ADA positive result at baseline for LAG525
Time Frame: Baseline
Population: LAG525 Immunogenicity (IG) prevalence set: all participants in the FAS wo received at least one dose of LAG525 with a determinant baseline LAG525 IG sample or at least one determinant post-baseline LAG525 IG sample.
Measure: Count of Participants; unit: Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 18 | 34 | 33
Participants | 0 | 0 | 1

24. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) on Treatment for LAG525
Description: Number of participants who were treatment-induced ADA positive for LAG525 (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive for LAG525 (post-baseline ADA positive with titer that was at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: From Cycle 1 to Cycle 7 (Day 1 pre-infusion) and end of treatment, assessed up to 3 years
Population: LAG525 immunogenicity incidence set: all participants in the LAG525 immunogenicity prevalence set with a determinant LAG525 baseline IG sample and at least one determinant LAG525 post-baseline IG sample.
Measure: Count of Participants; unit: Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 15 | 32 | 32
Participants | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) at Baseline for PDR001
Description: Number of participants who had an ADA positive result at baseline for PDR001.
Time Frame: Baseline
Population: PDR001 Immunogenicity (IG) prevalence set: all participants in the FAS who received at least one dose of PDR001 with a determinant baseline PDR001 IG sample or at least one determinant post-baseline PDR001 IG sample
Measure: Count of Participants; unit: Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 18 | 34
Participants | 3 | 6

26. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) on Treatment for PDR001
Description: Number of participants who were treatment-induced ADA positive for PDR001 (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive for PDR001 (post-baseline ADA positive with titer that was at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: From Cycle 1 to Cycle 7 (Day 1 pre-infusion) and end of treatment, assessed up to 2.8 years
Population: PDR001 Immunogenicity incidence set: all subjects in the PDR001 Immunogenicity prevalence set with a determinant PDR001 baseline IG sample and at least one determinant PDR001 post-baseline IG sample.
Measure: Count of Participants; unit: Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin
Number analyzed (Participants) | 15 | 25
Participants | 1 | 0

27. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after the last dose of study medication for a maximum duration of 2.9 years.
  Extended safety follow up deaths were collected from day 31 post treatment up to 150 days post-treatment, for a maximum duration of 3.2 years.
  Post-treatment deaths were collected after 150 days post-treatment, for a maximum duration of 3.2 years.
Time Frame: Up to 2.9 years (on-treatment), up to 3.2 years (extended safety follow-up and post-treatment)
Population: Safety set: all participants who received at least one dose of study treatment (i.e., at least one dose of any component of the study treatment, including incomplete infusion of spartalizumab, LAG525 or carboplatin).
Measure: Count of Participants; unit: Participants
Arm/Group | LAG525 + PDR001 | LAG525+ PDR001+ Carboplatin | LAG525 + Carboplatin
Number analyzed (Participants) | 19 | 34 | 34
Participants
  On-treatment | 0 | 2 | 1
  Extended safety follow-up deaths | 7 | 7 | 16
  Post-treatment deaths | 8 | 15 | 11
  All deaths | 15 | 24 | 28

ADVERSE EVENTS:
Time Frame: In the on-treatment period, adverse events (AEs) and serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to 2.9 years In the extended safety follow-up period, AEs and serious AEs (including the All-Cause Mortality data table) are presented from day 31 to day 150 after last administration of study treatment, up to 3.2 years
Description: The safety analysis was performed in the safety set including all participants who received at least one dose of study treatment (i.e., at least one dose of any component of the study treatment, including incomplete infusion of spartalizumab, LAG525 or carboplatin).
Groups:
- LAG525 + PDR001 (On-treatment Period); LAG525 + PDR001 (Extended Safety Follow-up Period): Participants received LAG525 and PDR001 administered as infusion once every 3 weeks
- LAG525 + PDR001+Carboplatin (On-treatment Period); LAG525 + PDR001+Carboplatin (Extended Safety Follow-up Period): Participants received LAG525, PDR001 and carboplatin administered as infusion once every 3 weeks.
- LAG525 +Carboplatin (On-treatment Period); LAG525 +Carboplatin (Extended Safety Follow-up Period): Participants received LAG525 and carboplatin administered as infusion once every 3 weeks
Arm/Group | LAG525 + PDR001 (On-treatment Period) | LAG525 + PDR001 (Extended Safety Follow-up Period) | LAG525 + PDR001+Carboplatin (On-treatment Period) | LAG525 + PDR001+Carboplatin (Extended Safety Follow-up Period) | LAG525 +Carboplatin (On-treatment Period) | LAG525 +Carboplatin (Extended Safety Follow-up Period)
All-Cause Mortality (participants affected / at risk) | 0/19 | 7/19 | 2/34 | 7/34 | 1/34 | 16/34
Serious Adverse Events (participants affected / at risk) | 6/19 | 0/19 | 12/34 | 6/34 | 14/34 | 2/34
Other Adverse Events (participants affected / at risk) | 17/19 | 0/19 | 34/34 | 11/34 | 33/34 | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAG525 + PDR001 (On-treatment Period) (N=19) | LAG525 + PDR001 (Extended Safety Follow-up Period) (N=19) | LAG525 + PDR001+Carboplatin (On-treatment Period) (N=34) | LAG525 + PDR001+Carboplatin (Extended Safety Follow-up Period) (N=34) | LAG525 +Carboplatin (On-treatment Period) (N=34) | LAG525 +Carboplatin (Extended Safety Follow-up Period) (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LAG525 + PDR001 (On-treatment Period) (N=19) | LAG525 + PDR001 (Extended Safety Follow-up Period) (N=19) | LAG525 + PDR001+Carboplatin (On-treatment Period) (N=34) | LAG525 + PDR001+Carboplatin (Extended Safety Follow-up Period) (N=34) | LAG525 +Carboplatin (On-treatment Period) (N=34) | LAG525 +Carboplatin (Extended Safety Follow-up Period) (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 20 | 5 | 19 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 1 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 15 | 0 | 14 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 5 | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 5 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 5 | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 7 | 1 | 16 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 5 | 2 | 7 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 18 | 2 | 13 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7 | 1 | 7 | 0
Asthenia (General disorders) | 0 | 0 | 11 | 0 | 5 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 11 | 1 | 12 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 2 | 0 | 2 | 0
Malaise (General disorders) | 1 | 0 | 3 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 4 | 0 | 3 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 6 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 4 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 4 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 11 | 2 | 6 | 0
Platelet count decreased (Investigations) | 1 | 0 | 14 | 2 | 9 | 0
SARS-CoV-2 test negative (Investigations) | 0 | 0 | 2 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 5 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 4 | 0 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 7 | 2 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 2 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 6 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 8 | 0 | 4 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 6 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 7 | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 6 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 6 | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03499899/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03499899/SAP_001.pdf